CLINICAL TRIAL: NCT00124072
Title: SEARCH: Study of the Effectiveness of Additional Reductions in Cholesterol and Homocysteine
Brief Title: Study of the Effectiveness of Additional Reductions in Cholesterol and Homocysteine
Acronym: SEARCH
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Professor Rory Collins, University of Oxford
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CTSUSEARCH1
Record Dates: First submitted 2005-07-22; First posted 2005-07-26 (Estimated); Results first posted 2010-06-09 (Estimated); Last update posted 2012-02-01 (Estimated); Status verified 2012-01

CONDITIONS: Cardiovascular Disease
Keywords: Myocardial infarction; Coronary heart disease; Cholesterol; Stroke
MeSH Terms: conditions — Cardiovascular Diseases; Myocardial Infarction; Coronary Disease; Stroke | interventions — Simvastatin; Folic Acid; Vitamin B 12

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Simvastatin 20 mg + folic acid and B12 (Active Comparator): Participants received 20 mg simvastatin once daily, and 2 mg folic acid with 1 mg vitamin B12 once daily
  Interventions: Drug: Simvastatin 20 mg daily; Dietary Supplement: Folic acid 2 mg + vitamin B12 1 mg daily
- Simvastatin 80 mg + folic acid and B12 (Active Comparator): Participants received 80 mg simvastatin once daily, and 2 mg folic acid with 1 mg vitamin B12 once daily
  Interventions: Dietary Supplement: Folic acid 2 mg + vitamin B12 1 mg daily; Drug: Simvastatin 80 mg daily
- Simvastatin 20 mg + placebo (Active Comparator): Participants received 20 mg simvastatin once daily, and placebo folic acid with placebo vitamin B12 once daily
  Interventions: Drug: Simvastatin 20 mg daily; Drug: Placebo
- Simvastatin 80 mg + placebo (Active Comparator): Participants received 80 mg simvastatin once daily, and placebo folic acid with placebo vitamin B12 once daily
  Interventions: Drug: Simvastatin 80 mg daily; Drug: Placebo

INTERVENTIONS:
Drug: Simvastatin 20 mg daily — Simvastatin 20 mg tablet once daily
  Arms: Simvastatin 20 mg + folic acid and B12; Simvastatin 20 mg + placebo
Dietary Supplement: Folic acid 2 mg + vitamin B12 1 mg daily — Folic acid 2 mg + vitamin B12 1 mg tablet once daily
  Arms: Simvastatin 20 mg + folic acid and B12; Simvastatin 80 mg + folic acid and B12
Drug: Simvastatin 80 mg daily — Simvastatin 80 mg tablet once daily
  Arms: Simvastatin 80 mg + folic acid and B12; Simvastatin 80 mg + placebo
Drug: Placebo — Placebo vitamin B12/folic acid tablet once daily
  Arms: Simvastatin 20 mg + placebo; Simvastatin 80 mg + placebo

SUMMARY:
SEARCH is a randomised, double-blind, multi-centre United Kingdom (UK) trial of 12,064 patients with myocardial infarction (MI) prior to study entry which aims to demonstrate whether a more intensive cholesterol lowering regimen using 80 mg simvastatin daily produces a larger and worthwhile reduction in cardiovascular events compared with a standard 20 mg daily regimen and whether reducing blood homocysteine levels with a daily dose of folic acid 2 mg + vitamin B12 1 mg compared with matching placebo produces a worthwhile reduction in vascular disease.

DETAILED DESCRIPTION:
In observational studies, lower blood cholesterol concentrations are associated with lower coronary risk, without any clear threshold below which lower levels are not associated with lower risk. Cholesterol reduction with statins reduces such risk but there is uncertainty about whether greater reductions with more intensive statin therapy will produce greater benefits. Elevated blood homocysteine levels appear to be an independent marker of cardiovascular risk, but it is unknown whether taking vitamins to reduce homocysteine concentrations will translate into cardiovascular benefit.

12,064 survivors of myocardial infarction have been randomised in a 2x2 factorial design to more intensive versus standard cholesterol-lowering treatment, using 80 mg or 20 mg daily simvastatin, and separately to homocysteine-lowering with folic acid plus vitamin B12 or matching placebo. Follow-up will continue until there are at least 2800 confirmed major vascular events (MVE), defined as non-fatal myocardial infarction, coronary death, stroke or arterial revascularisation. The primary outcome is the incidence of first MVE during the scheduled treatment period.

SEARCH should provide reliable evidence of the effectiveness and safety of more intensive cholesterol-lowering for the reduction of major vascular events in a high-risk population, and of the effects of homocysteine-lowering with folic acid plus vitamin B12.

ELIGIBILITY:
Inclusion Criteria:

* Prior myocardial infarction
* Statin therapy indicated
* No clear indication for folic acid

Exclusion Criteria:

* No clear contraindication to study treatments
* Screening plasma total cholesterol <3.5 mmol/l in patient already on statin therapy, or <4.5 mmol/l in patient not on statin therapy
* Chronic liver disease
* Severe renal disease or evidence of renal impairment
* Inflammatory muscle disease
* Concurrent treatment with fibrates or high-dose niacin
* Concurrent treatment with cyclosporin (or condition likely to result in organ transplantation and the need for cyclosporin), nefazodone, methotrexate, systemic azole antifungal or systemic macrolide antibiotics
* Child bearing potential
* No other predominant medical problem (other than coronary heart disease [CHD]) which might limit compliance with 5 years of study treatment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12064 (Actual)
Dates: Start 1998-07; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rory Collins, MB BS FRCP, Study Director — University of Oxford
Locations (1):
- CTSU, Richard Doll Building, University of Oxford, Oxford, Oxon, United Kingdom

REFERENCES:
- See also: SEARCH study website (primarily for dissemination of the results) — http://www.searchinfo.org/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First Patient In: 28-SEP-1998, Last Patient Last Visit: 22-May-2008 Eighty-eight (88) sites in 3 countries: England 72, Scotland 12 and Wales 4.
Pre-assignment Details: Patients entered a run-in period during which they received simvastatin 20 mg daily and placebo-vitamin tablets for 2 months. Eligible patients who completed run-in were then randomized in a 2x2 factorial blinded design between simvastatin 80 mg daily versus simvastatin 20 mg daily and folic acid 2 mg + vitamin B12 1 mg daily versus placebo.
Period: Overall Study
Arm/Group | Simvastatin 20 mg + Folic Acid and B12 | Simvastatin 80 mg + Folic Acid and B12 | Simvastatin 20 mg + Placebo | Simvastatin 80 mg + Placebo
Started | 3017 | 3016 | 3016 | 3015
Completed | 2503 | 2504 | 2524 | 2515
Not Completed | 514 | 512 | 492 | 500
Not completed — Lost to Follow-up for Mortality | 0 | 3 | 2 | 2
Not completed — Lost to Follow-up for Morbidity | 15 | 25 | 19 | 18
Not completed — Death | 499 | 484 | 471 | 480

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Simvastatin 20 mg + Folic Acid and B12 | Simvastatin 80 mg + Folic Acid and B12 | Simvastatin 20 mg + Placebo | Simvastatin 80 mg + Placebo | Total
Number analyzed (Participants) | 3017 | 3016 | 3016 | 3015 | 12064
Age Continuous [Mean (Standard Deviation); unit: years] | 64.2 (8.9) | 64.2 (8.9) | 64.2 (8.9) | 64.2 (8.9) | 64.2 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 513 | 514 | 513 | 512 | 2052
  Male | 2504 | 2502 | 2503 | 2503 | 10012
Region of Enrollment [Number; unit: participants]
  United Kingdom | 3017 | 3016 | 3016 | 3015 | 12064

OUTCOME MEASURES:

1. Primary Outcome: Major Vascular Events (MVE)
Description: Major vascular events (MVE) defined as major coronary events (MCE [non-fatal MI, coronary death or coronary revascularisation]), non-fatal or fatal stroke, or peripheral revascularization (peripheral artery angioplasty or arterial surgery, including amputations), during the scheduled study treatment period.
Time Frame: 6.7 years median follow-up
Measure: Number; unit: Participants
Groups:
- Simvastatin 20 mg Daily: Simvastatin 20 mg tablet once daily in the following arms: simvastatin 20 mg daily + folic acid 2 mg and vitamin B12 1 mg daily (active); simvastatin 20 mg daily + placebo vitamin B12/folic acid
- Simvastatin 80 mg Daily: Simvastatin 80 mg tablet once daily in the following arms: simvastatin 80 mg daily + folic acid 2 mg and vitamin B12 1 mg daily (active); simvastatin 80 mg daily + placebo vitamin B12/folic acid
- Folic Acid 2 mg + Vitamin B12 1 mg Daily: Folic acid 2 mg + vitamin B12 1 mg tablet once daily in the following arms: simvastatin 20 mg daily + folic acid 2 mg and vitamin B12 1 mg daily (active); simvastatin 80 mg daily + folic acid 2 mg and vitamin B12 1 mg daily (active)
- Placebo: Placebo vitamin B12/folic acid tablet once daily in the following arms: simvastatin 20 mg daily + placebo vitamin B12/folic acid; simvastatin 80 mg daily + placebo vitamin B12/folic acid
Arm/Group | Simvastatin 20 mg Daily | Simvastatin 80 mg Daily | Folic Acid 2 mg + Vitamin B12 1 mg Daily | Placebo
Number analyzed (Participants) | 6033 | 6031 | 6033 | 6031
Participants | 1553 | 1477 | 1537 | 1493

2. Secondary Outcome: MVEs Separately in Year 1 and in Later Years
Time Frame: 6.7 years median follow-up
Reporting Status: Not Posted
Measure: Number; unit: Participants

3. Secondary Outcome: MVEs in Patients Subdivided Into 3 Groups by Baseline Low-density Lipoprotein (LDL)
Time Frame: 6.7 years median follow-up
Reporting Status: Not Posted
Measure: Number; unit: Participants

4. Secondary Outcome: MVEs in Presence and Absence of the Other Factorial Treatment
Time Frame: 6.7 years median follow-up
Reporting Status: Not Posted
Measure: Number; unit: Participants

5. Secondary Outcome: Major Coronary Events
Description: Non-fatal MI, coronary death or coronary revascularisation
Time Frame: 6.7 years median follow-up
Reporting Status: Not Posted
Measure: Number; unit: Participants

6. Secondary Outcome: Total Strokes
Time Frame: 6.7 years median follow-up
Reporting Status: Not Posted
Measure: Number; unit: Participants

ADVERSE EVENTS:
Time Frame: 6.7 years median follow-up
Arm/Group | Simvastatin 20 mg Daily | Simvastatin 80 mg Daily | Folic Acid 2 mg + Vitamin B12 1 mg Daily | Placebo
Serious Adverse Events (participants affected / at risk) | 5037/6033 | 5024/6031 | 5068/6033 | 4993/6031
Other Adverse Events (participants affected / at risk) | 479/6033 | 493/6031 | 480/6033 | 492/6031
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Simvastatin 20 mg Daily (N=6033) | Simvastatin 80 mg Daily (N=6031) | Folic Acid 2 mg + Vitamin B12 1 mg Daily (N=6033) | Placebo (N=6031)
MVE (Vascular disorders) | 1553 | 1477 | 1537 | 1493
Other (General disorders) | 3484 | 3547 | 3531 | 3500
OTHER ADVERSE EVENTS (reported when occurring in more than 2.5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Simvastatin 20 mg Daily (N=6033) | Simvastatin 80 mg Daily (N=6031) | Folic Acid 2 mg + Vitamin B12 1 mg Daily (N=6033) | Placebo (N=6031)
Abdominal pain or indigestion (Gastrointestinal disorders) | 143 | 167 | 156 | 154
Tiredness or lethargy (General disorders) | 165 | 152 | 162 | 155
Other and unspecified symptom or problem (General disorders) | 171 | 174 | 162 | 183

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes